

The elderly patient demented in an acute geriatric department: pilot study, monocentric, randomized on the use of aromatherapy as a complementary treatment tool to psychopharmacology in behavioral and psycological symptoms of dementia (BPSD)

Protocol version: n.3, 23 of April 2018

Activation date: May 2018

NCT03662360

When 2 Of 32

### **INDEX**

| 1. | Synopsis | pag. 4 |
|-----|------------------------------------|---------|
| 2. | Flow chart | pag. 7 |
| 3. | Study characteristics | pag. 9 |
| 4. | Protocol rationale | pag. 9 |
| 5. | Study population | pag. 10 |
| 6. | Project objectives | pag. 12 |
| 7. | Randomization | pag. 13 |
| 8. | Project design | pag. 13 |
| 9. | Eligibility criteria | pag. 15 |
| 10. | Codify and registration procedures | pag. 15 |
| 11. | Project duration | pag. 15 |
| 12. | Risks and benefits | pag. 15 |
| 13. | Statistical considerations | pag. 16 |
| 14. | Ethical considerations | pag. 16 |
| 15. | Data publishing policy | pag. 16 |
| 16. | Insurance coverage | pag. 16 |
| 17. | Funding | pag. 16 |
| 18. | Conflicts of interest | pag. 16 |
| 19. | Additional information | pag. 16 |
| 20. | Bibliography | pag. 17 |
| 21. | Appendix | pag. 20 |
| | 21.1 Scores used for evaluation | pag. 20 |

Version No.3 of 23.04.2018 When 3 Of 32

#### 1. SYNOPSIS

The elderly patient demented in an acute geriatric department: pilot study, monocentric, randomized on the use of aromatherapy as a complementary treatment tool to psychopharmacology in psychological disorders and behavior (BPSD).

#### Rationale

Behavioral and psycological symptoms of dementia (BPSD) are a big issue for families, paramedics, physician and the patient itself (1,2,3,4).

In absence of universally recognized guidelines, the standard of treatment of these disorders involves the use of psychotropic drugs (typical/atypical neuroleptics, antidepressants, benzodiazepines) that are often found to have a reduce efficacy and induce a number of side effects such as sedation, impaired motor neurons slowdown, cardiac electrical alterations and extrapyramidal syndrome (5,6,7,8,9). In consideration of this, it is important to check for treating alternative ways, which can reduce psychological and behavioural disorders and at the same time can reduce the use of psychotropic drugs.

Concerning the aromatherapy [10], the therapeutic use of natural essential oils, there are decades of clinical experience, especially in France, accompanied by increasing scientific evidence with significant increase in publications regarding its use of psychological disorders and dementiarelated behavior context (11,12,13,14).

Based on the available scientific publications, it has been therefore decided to use two essential oils (*Citrus sinensis*, *Lavandula angustifolia*) in environmental diffusion within the Geriatric Department of the Clinic Luganese Moncucco.

#### **Objectives**

Primary objectives: through the execution of the Neuropsychiatric Inventory — Nursing Home Version (NPI-NH), the neuropsychiatric and psychopathological symptoms of dementia patients will be evaluated in order to assess how the use of aromatherapy can improve the management of BPSD, reducing, where there is clinical indication, psychotropic therapy and secondary side effects. The score is considered positive if the presence of BPSD is greater than or equal to 1 (15, 16,17); the improvement of the score is represented from decrease of the NPI-NH respect to the initial assessment (19, 20). Performing neuropsychological tests is not an additional attention to enrolled patients, but it is part of clinical practice (18).

Secondary objectives: to validate the hypothesis that through the use of aromatherapy will improved the management of Behavioral and psycological symptoms of dementia (BPSD) in the dementia patient, with a concomitant reduction of the clinical staff stress who take care of patients (physician, nurses, care assistants), determined by the results reported by the Neuropsychiatric Inventory – Nursing Home Version (NPI-NH), In the specific section concerning

the distress measurement; improvement of the score is represented from decrease of the NPI-NH respect to the initial assessment (19, 20).

Project duration: 2 months of enrollment.

**Number of patients:** 32, 16 patients for the control group and 16 patients for the group" aromatherapy".

#### Inclusion criteria:

- patients age ≥ 70 years;
- patients admitted to the acute geriatrics ward;
- patients with known diagnosis of dementia associated with BPSD or diagnosis performed during hospitalization.

#### **Exclusion criteria:**

- patients with alcohol-based dementia;
- patients with Mild Cognitive Impairment (MCI) paragraph 4;
- patients with language barriers;
- patients already being treated with aromatherapy.

**Protocol design:** prospective data collection of psychological disorders and behaviour in patients with diagnosis of dementia with associated behavioral and psycological symptoms of dementia (BPSD)- diagnosis already performed using neuropsychological tests (below), according Evidence Based Medicine, and/or patients who BPSD diagnosis performed during the hospital stay in the Geriatric Competence Centre, Clinica Luganese Moncucco.

The enrollment will be performed in May and June 2018.

Enrolled patients will be treated with psychotropic drugs vs psychotropic drugs with aromatherapy in environmental diffusion. It is expected to use neuropsychological specific tests to assess dementia, motor and functional status patient status (CAM - Confusion Assessment Method -, CDR - Clinical Dementia Rating -, MMSE - Mini Mental State Examination -, FAB - Frontal Assessment Battery -, Tinetti Scale, BADL - Basic Activities of Daily Living -, IADL - Instrumental Activities of Daily Living -, NPI-NH — Neuropsychiatric Inventory — Nursing Home Version)).

Patients enrolled in the project will not undergo to additional tests; the performed test are required in the standard clinical practice [18].

**GROUP A:** 16 patients, following the inclusion criteria, will be enroll and they will be treated with psychotropic drugs.

**GROUP B:** 16 patients, following the inclusion criteria, will be enroll and they will be treated with psychotropic drugs and, in a complementary way, with aromatherapy in environmental diffusion.

# 2. FLOW CHART Patients hospitalized in the acute geriatric dept from May to June 2018 Inclusion criteria: Exclusion criteria: - patients ≥ 70 years; - patients with alcohol-based dementia; - patients admitted to the Acute Geriatric - patients with Mild Cognitive Impairment Ward: (MCI); - patients with BPSD; - patients with language barriers; - patients already treated with aromatherapy. Patients enrollment (T0) Signature of **Informed Consent Form Acceptance** Non-acceptance Randomization in Group A or B **Observation** for 48 hrs an data collection: - age: - male or female; - CAM (Confusion Assessment Method); - CDR (Clinical Dementia Rating Score) - MMSE (Mini Mental State Examination); - FAB (Frontal Assessment Battery); - Tinetti's scale; - BADL (Basic Activities of Daily Living); - IADL (Instrumental Activities of Daily Living); - number/types of neuroleptics; - number/types of antidepressants; - number/types of benzodiazepines. **NPI-NH** rating: - NPI physician; - NPI nurse: - NPI care assistant. If NPI-NH >/= 1 If NPI = 0

Version No.3 of 23.04.2018 When 7 Of 32



Version No.3 of 23.04.2018 When 8 Of 32

#### 3. STUDY CHARACTERISTIC

Monocentric, randomized, pilot study which consists in the prospective data collection related to psychological disorders and behavior in the patient with dementia using neuropsychological tests in order to define the possible effectiveness of two essential oils (*Citrus sinensis*, *Lavandula angustifolia*) in the disorders control of psychological sphere and behavior of patients with degenerative or mixed type of dementia, admitted in the Geriatric Department of Clinica Luganese Moncucco in May and June 2018.

In the proposal for therapeutic process of dementia patients in this project there is no disaccording with Evidence Based Medicine.

Patients enrolled in the project will not undergo additional tests; the performed tests will follow the standard procedures of clinical practice [18].

#### 4. PROTOCOL RATIONALE

Behavioral and psycological symptoms of dementia (BPSD) are a major problem for families, physicians and the patient itself [1,2,3,4].

Performing neuropsychological tests is not an additional source of distress for enlisted patients, but is part of clinical practice [18].

The standard treatment of these disorders involves the use of psychotropic drugs (typical/atypical neuroleptics, antidepressants, benzodiazepines) which are often ineffective and have a number of side effects such as sedation, reduction in cognitive performance, cardiac electrical alterations and extrapyramidal syndrome [5,6,7,8,9].

Within the scientific community, it is therefore mandatory to identify alternative ways of managing BPSDs, which can have a beneficial effect on patient life and, at the same time, a reduction in the used of psychotropic drugs.

The therapeutic use of natural essential oils has decades of clinical experience, especially in France, accompanied by an increase numbers of publications in their use in BPSD [11,12,13,14].

The knowledge of alternative treatments of BPSD (such as aromatherapy) are the basis of our study project, which involves the introduction of essential oils in the BPSD management, while maintaining conventional psychotropic therapy (typical/atypical neuroleptics, antidepressants, benzodiazepines) in a prefixed form of ProReNata (PRN) (paragraph 5).

The identified oils (*Citrus sinensis, Lavender angustifolia*) were selected on the degree of purity defined by the mass spectrophotometry available by the supplier.999

The choice of adjuvant therapy with essential oils could allow, in accordance with the 3rd principle of Medical Ethics to administer natural treatment to patients with distress with BPSD reducing, if possible, use of psychotropic drugs and their major side effects.

The use of essential oils in treatment of BPSD can also have a positive impact on patient economic management due to limited costs, allowing a distribution of treatments according to IV Principle of Ethics Medical: principle of justice.

Mild Cognitive Impairment (MCI) patients were excluded from the protocol as a form of predementia.[21].

MCI is a neurological syndrome characterized by a cognitive impairment greater than that statistically expected based on age and education level, but who are still able to carry out their daily activities (BADL and IADL tests). The Mild Cognitive Impairment is considered a form of predementia, situated in a transition point between normal aging and dementia.

#### 5. STUDY POPULATION

The population that will be evaluated within the project is constitute by patients with diagnosed dementia with BPSD (diagnosis carried out using, according to Evidence Based Medicine, the neuropsychological tests below) and/or by patients who the diagnosis of dementia with BPSD will be performed at the Geriatric Competence Centre of the Clinica Luganese Moncucco.

The enrollment will be performed in May and June 2018.

All patients mentioned above, within 48 hours after the admission at the Geriatric Department or the manifestation of BPSD, will be assessed to neuropsychological and functional tests (CAM - Confusion Assessment Method -, CDR - Clinical Dementia Rating Score -, MMSE - Mini Mental State Examination -, FAB - Frontal Assessment Battery -, scala di Tinetti, BADL - Basic Activities of Daily Living -, IADL - Instrumental Activities of Daily Living -), as required by Good Clinical Practice[18]. Subsequently, patients who can be enrolled in the study will be randomized into two groups, described below.

Here is the study population on which we will focus:

**GROUP A – controls** -: will be enrolled 16 patients eligible for criteria of inclusion, treated with psychotropic drugs.

**GROUP B – aromatherapy –:** will be enrolled 16 patients eligible for criteria of inclusion, treated with psychotropic drugs and aromatherapy in air-diffusion.

Based on the randomization, patients will be divided into group A – controls – and group B – aromatherapy in air diffusion.

Neuropsychiatric Inventory (NPI) is a validated and useful tool for characterizing and assessing the BPSD frequency and seriousness.

A Resident Physician will perform the NPI in our study protocol.

The physician, by interview with patient's nurse, in absence of patient himself, will fill out the NPI-NH.

The above mentioned physician, formerly operating in the Geriatric Department – who knows the geriatric assessments - and currently active in the Rheumatology Department, will therefore respect the blind study procedure.

The geriatric nurse was chosen for the close relationship of care that is created with the patient; during the test, BPSD frequency and seriousness will be evaluated.

The psychological distress induced by BPSD patients, will be evaluated on the three figures who have in charge the patient, which are nurses, care assistants and the resident physicians.

The psychological distress assessment is part of the NPI-NH test with a scale of severity from 0 to 5.

Nurses will be undergo to NPI – NH test within 48 hours after patient admission or at first appearance of BPSD (T1), T2 (T1-3 days) 3 days after enrollment, at T3 (T1-6 days) 6 days after enrollment, at T4 (T1-12 days) at 14th day. According to the same timing, NPI-NH will also be performed to the resident physicians, the nurses and the care assistants to assess the psychological distress. The NPI-NH test will be performed following the Good Clinical Practice.

The tests results performed to the two groups of patients will be considered in order to assess a possible reduction in BPSD. As the project is a pilot study, a descriptive analysis will be performed.

Here the schemes defined for treatment with aromatherapy and psychotropic drugs, according to scientific publications in the first case and scientific publications and Evidence Based Medicine in the second:

#### **Aromatherapy**

Route of administration: air diffusion with ultrasonic diffuser in a single room and for about an hour.

#### Doses:

- Citrus sinensis: 6 drops at 8, 12 and 18 in nebulization

and

- Lavender angustifolia: 6 drops 8 p.m. in nebulization

#### PRN PSYCOPHARMACOTHERAPY

#### Drug:

- in case of psychomotor agitation:

Haloperidol 1 mg PO 10 times in 24 hours

1 mg SC/IM 5 times in 24 hours

Reperidone 0.5mg - 2mg PO in 24 hours

Olanzapine 2.5 mg - 5 mg PO in 24 hours

Clozapine 6.25 mg – 25 mg PO in 24 hours

Version No.3 of 23.04.2018 When 11 Of 32

Quetiapine 12.5mg - 150mg PO in 24 hours

- in case of sleep disturbance:

Valerian 1 tb - 2 tbs PO in 24 hours

Melatonin 1 tb - 2 tbs PO in 24 hours

Lorazepam 0.5 mg - 3mg PO in 24 hours

Oxazepam 7.5mg - 45mg PO in 24 hours

Clomethiazole 1 tb -3 tbs PO in 24 hours

- in case of anxiety/depression:

Trazodone 25 mg – 150 mg PO in 24 hours

Escitalopram 10 mg - 20 mg PO in 24 hours

Mirtazapine 15 mg - 45 mg PO in 24 hours

Citalopram 10 mg - 20 mg PO in 24 hours

Paroxetine 20 mg – 50 mg PO in 24 hours

The control group is treated with psychopharmacological therapy, defined by the PI, according to the Evidence Based Medicine criteria.

Patient can withdraw the ICF at any time.

The investigators could decide to withdraw a patient for safety and health.

The withdrawn patients will not be evaluated unless they have been treated for 8 days, useful to evaluate the aromatherapy efficacy.

In bibliography reported that essential oils in air diffusion are effective in 3 days. Additional 5 days of treatment allow to stabilize patient's condition and collect, through the NPI-NH test, changing in BPSD data.

Withdrawn patients will be followed according to the standards of care provided by the Clinica Luganese Moncucco.

#### 6. PROJECT OBJECTIVES

The goal of this project is to evaluate the effectiveness of aromatherapy in air diffusion in addition to psychotropic drugs in order to evaluate a possible reduction in BPSD.

The project's hypothesis is that GROUP B patients show an improvement in their BPSD. The performed neuropsychological tests will provide the answer to the project hypotesis.

**Primary objectives**: validate the hypothesis that the use of aromatherapy in air diffusion can improve the BPSD management, allowing a reduce in psychotropic therapy prescribed and its secondary side effects. The patient's nurses will be tested with NPI-NH, that will characterize

frequency and seriousness of BPSD [15,16, 17]. A score greater or equal to 1 is considered positive for presence of BPSD.

**Secondary objectives**: validate the hypothesis that the use of aromatherapy will improve the management of BPSD patients, with a simultaneously reduction of physicians, nurses and care assistants stress. The last aspect will be evaluated with a specific part of NPI-NH test. The decrease of the initial score represented an improvement [19.20]. The NPI-NH test will be performed according to the time points defined in paragraph 7.1.1

The obtained results could be interesting to the future implementation of the use of essential oils in air diffusion in acute geriatric departments and in all facilities with BPSD patients.

#### 7. RANDOMIZATION

Enrolled patients with BPSD will be randomized according to the following randomization scheme (AABB, ABAB, BBAA, BABA, BABA, BAAB).

A repetition of the first 4blocks will be performed, for a total of 32 patients, 16 each group, according to the following scheme:

AABB, ABAB, BBAA, BABA AABB, ABAB, BBAA, BABA

#### 8. PROJECT DESIGN

The project will be managed in the acute geriatric department of the Clinica Luganese Moncucco. Enrolment and treatment scheme is present in the flow chart (chapter 2).

After randomization patients will be enrolled in the two groups GROUP A, control group, and GROUP B, treatment group.

The enrollment will be performed in 2 months.

**GROUP A:** 16 patients, following the inclusion criteria, will be enroll and they will be treated with psychotropic drugs.

**GROUP B:** 16 patients, following the inclusion criteria, will be enroll and they will be treated with psychotropic drugs and, in a complementary way, with aromatherapy in environmental diffusion.

The project hypothesis will be validated using the following neuropsychological and functional tests:

- CAM (Confusion Assessment Method);
- CDR (Clinical Dementia Rating Score)
- MMSE (Mini Mental State Examination);
- FAB (Frontal Assessment Battery);

- Tinetti's scale;
- BADL (Basic Activities of Daily Living);
- IADL (Instrumental Activities of Daily Living);
- NPI-NH (Neuropsychiatric Inventory Nursing Home Version);

Neuropsychological tests are part of clinical practice [18].

Scientific reports show that essential oils in air diffusion are effective in 3 days. A final timepoints of 14 days represent the mean hospital stay:

2 days for the collection of behavioral data;

6 days to observe the possible effectiveness of aromatherapy in air diffusion;

6 days to adapt the therapy with oils and psychotropic drugs and stabilize patient's condition for a possible discharge.

Enrolled patients and nurses will be tested according to the following times:

- **8.1.1 Observation for 48 hours with data collection and execution of the NPI-NH (T1)**: in the 48 hours after patient admission at the Geriatric Department or at the diagnosis of dementia, the information collection will be performed: sensitive data (age, gender), dementia condition (CAM, CDR, MMSE, FAB), functional status (IADL, BADL, Tinetti scale) and the used number of psychotropic drugs. As a result of this evaluation, patient will be assessed for the presence of BPSD using the NPI-NH assessment scale, nurses will be undergo to NPI NH test within 48 hours after patient admission. In case of a score greater than or equal to 1, patient will be followed within the study project, otherwise it will follow the standard process.
- **8.1.2** Assessment of NPI-NH at T2 (T1-3 days): 3 days after enrollment, patient will be re-evaluated with NPI-NH to assess BPSD progress. In addition, the distress level of on the three health caregivers is also measured with the NPI-NH test.
- **8.1.3** Assessment of NPI-NH at T3, assessment of vital parameters and use of drug reserves (T1-6 days): 6 days after enrollment, NPI-NH will be re-executed, with associated assessment of patient's vital signs (PAS, PAM, FC) and the use of psychotropic drug reserves.
- **8.1.4 Final T4 assessment (T1-12 days):** NPI-NH scale will be performed in association with vital signs.

The physician in charge of dispensing the NPI-NH questionnaires to nurses to collect BPSD patients status, will also submit the questionnaires to the referring physician, nurse and care assistants with the aim to assess the level of stress in the clinical staff (see "Distress" column in NPI-NH questionnaire in the appendix).

#### 9. ELEGIBILITY CRITERIA

#### Inclusion criteria:

- patients ≥ 70 years;
- patients admitted to the Acute Geriatric Ward;
- patients with known diagnosis of dementia associated with BPSD or diagnosis performed during the hospitalization.

#### **Exclusion criteria:**

- patients with alcohol-based dementia;
- patients with Mild Cognitive Impairment (MCI) paragraph 4 -;
- patients with language barriers;
- patients already being treated with aromatherapy.

Patients admitted to the Geriatric Competence Centre of the Clinica Luganese Moncucco who do not respect inclusion criteria at the time of admission but develop them in the course of stay in the Clinic (for example: patient without psychological disorders and behavior at the entrance that manifest BPSD during hospitalization) could be enrolled.

#### **10. CODIFY AND REGISTRATION PROCEDURES**

A unique and increasing patient number (UPN) will be assigned to each patient. The clinical research unit of Clinica Luganese Moncucco will keep the dataset containing the correspondence between the UPN and the patient's personal and clinical data. All the analyzed data, available for scientific discussions or publishing, will be encoded.

#### 11. PROJECT DURATION

Patients enrolment will be performed during May and June 2018.

#### 12. RISKS AND BENEFITS

This project involves the use of essential oils, which are natural and with no collateral risks; the only risks the patient might present are hypersensitivity to essential oil [22].

If aromatherapy results efficacious in the management of BPSD, patients benefit would result in a reduction of the use of psychotropic therapy with a consecutive reduction in the side effects.

At the same time as the effectiveness of aromatherapy, possible benefits will also be available for caregivers (doctors, nurses, patient care assistant, family members).

#### 13. STATISTICAL CONSIDERATIONS

This is a pilot study which required the enrollment of 32 patients. For this reason, the statistical considerations will be purely descriptive.

Patients will be enrolled, according to the described randomization, in GROUP A, control group in which patients will be treated exclusively with traditional psychotropics drugs, or in group B, in which they will be treated with aromatherapy integrated with psychotropics drugs.

#### **14.ETHICS CONSIDERATIONS**

This protocol has been designed and written in accordance with the Helsinki Agreement, the International Good Clinical Practice ICH Guidelines and the arrangements of the European and Swiss regulatory authorities [23, 24, 25].

In consideration of the presence of potentially vulnerable subjects, in order to ensure the inalienable principle of patient autonomy (I principle of Medical Ethics), informed consent will be explained and requested to a relative/legal representative of the patient who has lost the ability to discern.

#### 15. DATA PUBLISHING POLICY

The ownership of the data is of Clinica Luganese Moncucco. The results are also expected to be published in the event of negative results and the authors of the scientific work will be chosen according to their contribution.

#### **16. INSURANCE COVERAGE**

No specific insurance coverage is required.

#### 17. FUNDING

The funding for this pilot project comes from the aromatherapy fund of the Geriatric Competence Centre of Clinica Luganese Moncucco. This fund is funded by private donations. No companies participated in the financing.

#### **18. CONFLICTS OF INTEREST**

The authors and collaborators of the study declare that they do not present any conflict of interest.

#### 19. ADDITIONAL INFORMATION

As agreed with the Cantonal Ethics Committee, in order not to harm the sensitivity of patients and relatives involved in the study, the title of the protocol was changed only in informed consents, replacing the term "demented" with "with dementia." This measure has also not been applied to the protocol as it is a document that is not provided to relatives or involved patients, but is tool for the staff participating an the study.

#### **20. BIBLIOGRAPHY**

- 1. C.G. Ballard, S. Gauthier, J.L. Cummings et al. *Management of agitation and aggression associated with Alzheimer disease*. Nature Reviews Neurology, vol. 5, no.5, pp. 245-255, 2009.
- 2. M. Marganallo-Lana, A. Swann, J. O'Brien et al. *Prevalence and pharmacological management of behavioural and psychological symptoms amongst dementia sufferers linving in care environment.* International Journal of Geriatric Psychiatry, vol. 16, no. 1, pp. 39-44, 2001.
- 3. E. Lonergan, J. Luxenberg, J. Colford. *Haloperidol for agitation in dementia*. The Cochrane Database of Systematic Reviews, no.2, Article ID CD002852, 2002.
- 4. C. Ballard and A. Corbett. *Agitation and aggression in people with Alzheimer's disease*. Current opinion in Psychiatry, vol. 26, no. 3, pp. 252-259, 2013.
- 5. C. Ballard and R. Howard. *Neuroleptic drugs in dementia: benefits and harm.* Nature Reviews Neuroscience, vol. 7, no. 6, pp. 492-500, 2006.
- 6. L.S. Schneider, K. Dagerman, P.S. Insel. *Efficacy and adverse effects of atypical antipsychotics for dementia: metanalysis of randomized, placebo-controlled trials.* The American Journal of Geriatric Psychiatry, vol.14, no.3, pp 191-210, 2006.
- 7. L.S. Schneider, P.N. Tariot, K.S. Dagerman et al. *Effectiveness of atypical antipsychotic drugs in patients with Alzheimer's disease.* The New England Journal of Medicine, vol.355, no.15, pp.1525-1538, 2006.
- 8. FDA Public Health Advisory. *Deaths with antipsychotics in elderly patients with behavioral disturbances*. 2005. https://www.fda.gov/Drugs/Drugsafety/ucm053171.htm.
- 9. C. Ballard, M.L. Hanney, M. Theodoulou et al. *The dementia antipsychotic withdrawal trial* (DART-AD): long-term follow-up of a randomised placebo-controlled trial. The Lancet Neurology, vol.8, no.2, pp.151-157, 2009.
- 10. C. Bagetta, M. Cosentino, T. Sakurada. *Preface in Aromatherapy: Basic Mechanisms and Evidence Based Clinical Use.* Oxfordshire, UK, Taylor & Francis, 2016.
- 11. C.G. Ballard, J.T. O'Brien, K.Reichelt, E.K. Perry. *Aromatherapy as a safe and effective treatment for the management of agitation in severe dementia: the results of a double-blind, placebo-controlled trial with Melissa*. Journal of Clinical Psychiatry, vol.63, no.7, pp.553-558, 2002.
- 12. C. Holmes, V. Hopkins, C. Hensford, V. MacLaughlin, D. Wilkinson, H. Rosenvinge. *Lavender oil as a treatment for agitated behaviour in severe dementia: a placebo controlled study*. International Journal of Geriatric Psychiatry, vol.17, no.4, pp.305-308, 2002.
- 13. D.W. O'Connor, B. Eppingstall, J. Taffe, E.S. Van Der Ploeg. *A randomized, controlled cross-over trial of dermally-applied lavender (Lavandula angustifolia) oil as a treatment of agitated behaviour in dementia*. BMC Complementary and Alternative Medicine, vol.13, article 315, 2013.

- 14. D. Jimbo, Y. Kimura. M. Taniguchi, M. Inoue, K. Urakami. *Effect of aromatherapy on patients with Alzheimer's disease*. Psychogeriatrics, vol.9, no.4, pp.173-179, 2009.
- E. Elisabetsky, J. Marschner, D. Onofre Souza. *Effects of linalool on glutamatergic system in the rat cerebral cortex.* Neurochemical Research, vol.20, no.4, pp.461-465, 1995.
- L. Huang, S. Abuhamdah, M.J.R. Howes et al. *Pharmacological profile of essential oils derived from Lavandula angustifolia and Melissa officinalis with anti-agitation properties: focus on ligand-gated channel.* Journal of Pharmacy and Pharmacology, vol.60, no.11, pp.1515-1522, 2008.
- J.T. Kim, C.J. Ren, G.A. Fielding et al. *Treatment with lavender aromatherapy in the post-anesthesia* care unit reduces opioid requirements of morbidly obese patients undergoing laparoscopic adjustable gastric banding. Obesity Surgery, vol.17, no.7, pp.920-925, 2007.
- E. Barocelli, F.Calcina, M. Chiavarini et al. *Antinociceptive and gastroprotective effects of inhaled and orally administered Lavandula Hybrida Reverchon "grosso" essential oil.* Lige Sciences, vol.76, no.2, pp.213-223, 2004.
- 15. Cummings JL. *The Neuropsychiatric Inventory: Assessing psychopathology in dementia patients*. Neurology 1997; 48 (Supple 6): S10-S16.
- 16. Cummings JL et al. *The Neuropsychiatric Inventory: comprenhensive assessment of psychopathology in dementia.* Neurology 1994; 44: 2308-2314.
- 17. Martini De Oliveira A et al. *Nonpharmacological Interventions to Reduce Behavioral and Psychological Symptoms of Dementia: A Systematic Review.* BioMed Research International 2015.
- 18. Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, Conroy SP, Kircher T, Somme D, Saltvedt I, Wald H, O'Neill D, Robinson D, Shepperd S. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. Sep 12;9, 2017
- 19. Kaufer DI et al. Assessing the impact of neuropsychiatric symptoms in Alzheimer's disease: the Neuropsychiatric Inventory caregiver Distress Scale. J Am Geriatr Soc 1998; 46: 210-215.
- 20. Wood S et al. The use of the Neuropsychiatric Inventory in nursing home residents, characterization and measurement. Am J Geriatr Psychiatry 2000; 8: 75-83.
- 21. <a href="https://www.uptodate.com/contents/mild-cognitive-impairment-epidemiology-pathology-and-clinical-assessment?search=mild%20cognitive%20impairment&source=search\_result&selectedTitle=1~15</a>
  0&usage type=default &display rank=1
- 22. Gyorgyi P et al. *Contact Hypersensitivity to Lavender Oil in Hungary: a Multicentre Survey 2013-2014*. Journal of dermartological research and therapy 2015; 1:26-32

- 23. Directive 2001/20/EC of the European Parliament and of the Council of 4 April 2001 on the approximation of the laws, regulations and administrative provisions of the member states relating to the implementation of good clinical practice in the conduct of clinical trials on medicinal products for human use. Medicinska etika a bioetika: casopis Ustavu medicinskej etiky a bioetiky = Medical ethics & bioethics: journal of the Institute of Medical Ethics & Bioethics. 2002; 9:12-9.
- 24. Dixon JR, Jr. The International Conference on Harmonization Good Clinical Practice Guideline (1998). Quality assurance; 6:65-74.
- 25. The Helsinki Declaration of the World Medical Association (WMA). Ethical principles of medical research involving human subjects]. Polski merkuriusz lekarski : organ Polskiego Medical Society. 2014; 36:298-301.

#### 21.APPENDIX

#### 21.1 Scores used for evaluation

## 21.1.1 Confusion Assessment Method (CAM)

| Confusion Assessment Method (CAM) | Date of assessment | | |
|---|---|---|---|
| Diagnostic Algorithm | Time of assessment | | |
| | | Yes or No | |
| Acute onset and fluctuating course? (Acute change i baseline, fluctuating behaviour through the day) | n mental status from | | |
| Inattention? (Difficulty focusing attention, easily distrack of what is being said) | | | |
| Disorganised thinking? (disorganized or incoherent the irrelevant conversation, unclear or illogical flow of ideas | | | |
| 4. Altered level of consciousness? (This feature is show "alert", including: hyper-alert, lethargic, stupor, or coma | | | |
| The diagnosis of Delirium by CAM requires the pres | ID EITHER 3 | or 4 | |
| Delirium detected? | | YES<br>(Circle) | NO |

Reference: Inouye SK, Van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI (1990) Clarifying confusion: the Confusion Assessment Method. *Annals of Internal Medicine* 113: 941-8

# 21.1.2 Mini Mental State Evaluation (MMSE)

# Mini-Mental State Examination (MMSE)

| Patient's Name: | Date: |
|-----------------|-------|

Instructions: Score one point for each correct response within each question or activity.

| Maximum<br>Score | Patient's<br>Score | Questions |
|---|---|---|
| 5 | | "What is the year? Season? Date? Day? Month?" |
| 5 | | "Where are we now? State? County? Town/city? Hospital? Floor?" |
| 3 | | The examiner names three unrelated objects clearly and slowly, then the instructor asks the patient to name all three of them. The patient's response is used for scoring. The examiner repeats them until patient learns all of them, if possible. |
| 5 | | "I would like you to count backward from 100 by sevens." (93, 86, 79, 72, 65,) Alternative: "Spell WORLD backwards." (D-L-R-O-W) |
| 3 | | "Earlier I told you the names of three things. Can you tell me what those were?" |
| 2 | | Show the patient two simple objects, such as a wristwatch and a pencil, and ask the patient to name them. |
| 1 | | "Repeat the phrase: 'No ifs, ands, or buts.'" |
| 3 | | "Take the paper in your right hand, fold it in half, and put it on the floor." (The examiner gives the patient a piece of blank paper.) |
| 1 | | "Please read this and do what it says." (Written instruction is "Close your eyes.") |
| 1 | | "Make up and write a sentence about anything." (This sentence must contain a noun and a verb.) |
| 1 | | "Please copy this picture." (The examiner gives the patient a blank piece of paper and asks him/her to draw the symbol below. All 10 angles must be present and two must intersect.) |
| 30 | | TOTAL |

## Interpretation of the MMSE:

| Method | Score | Interpretation |
|---------------|-------|----------------------------------------------|
| Single Cutoff | <24 | Abnormal |
| Range | <21 | Increased odds of dementia |
| Range | >25 | Decreased odds of dementia |
| | 21 | Abnormal for 8 <sup>th</sup> grade education |
| Education | <23 | Abnormal for high school education |
| | <24 | Abnormal for college education |
| | 24-30 | No cognitive impairment |
| Severity | 18-23 | Mild cognitive impairment |
| | 0-17 | Severe cognitive impairment |

#### Interpretation of MMSE Scores:

| Score | Degree of<br>Impairment | Formal Psychometric<br>Assessment | Day-to-Day Functioning |
|---|---|---|---|
| 25-30 | Questionably<br>significant | If clinical signs of cognitive impairment<br>are present, formal assessment of<br>cognition may be valuable. | May have clinically significant but mild deficits. Likely to affect only most demanding activities of daily living. |
| 20-25 | Mild | Formal assessment may be helpful to<br>better determine pattern and extent of<br>deficits. | Significant effect. May require some<br>supervision, support and assistance. |
| 10-20 | Moderate | Formal assessment may be helpful if there are specific clinical indications. | Clear impairment. May require 24-hour supervision. |
| 0-10 | Severe | Patient not likely to be testable. | Marked impairment. Likely to require<br>24-hour supervision and assistance<br>with ADL. |

Source:

• Folstein MF, Folstein SE, McHugh PR: "Mini-mental state: A practical method for grading the cognitive state of patients for the clinician." J Psychiatr Res 1975;12:189-198.

#### 21.1.3 Frontal Assessment Battery (FAB)

#### Frontal Assessment Battery

#### Purpose

The FAB is a brief tool that can be used at the bedside or in a clinic setting to assist in discriminating between dementias with a frontal dysexecutive phenotype and Dementia of Alzheimer's Type (DAT). The FAB has validity in distinguishing Fronto-temporal type dementia from DAT in mildly demented patients (MMSE > 24). Total score is from a maximum of 18, higher scores indicating better performance.

#### 1. Similarities (conceptualization)

"In what way are they alike?"

A banana and an orange

(In the event of total failure: "they are not alike" or partial failure: "both have peel," help the patient by saying: "both a banana and an orange are fruit"; but credit 0 for the item; do not help the patient for the two following items)

- A table and a chair
- A tulip, a rose and a daisy

Score (only category responses [fruits, furniture, flowers] are considered correct)

Three correct: 3 Two correct: 2 One correct: 1 None correct: 0

#### 2. Lexical fluency (mental flexibility)

"Say as many words as you can beginning with the letter 'S,' any words except surnames or proper nouns."

If the patient gives no response during the first 5 seconds, say: "for instance, snake." If the patient pauses 10 seconds, stimulate him by saying: "any word beginning with the letter 'S.' The time allowed is 60 seconds.

Score (word repetitions or variations [shoe, shoemaker], surnames, or proper nouns are not counted as correct responses)

> 9 words: 3 6 -9 words: 2 3 -5 words: 1 < 3 words: 0

#### 3. Motor series "Luria" test (programming)

"Look carefully at what I'm doing."

The examiner, seated in front of the patient, performs alone three times with his left hand the series of "fist-edge-palm."

"Now, with your right hand do the same series, first with me, then alone."

The examiner performs the series three times with the patient, then says to him/her:

"Now, do it on your own."

#### Score

Patient performs six correct consecutive series alone: 3
Patient performs at least three correct consecutive series alone: 2
Patient fails alone, but performs three correct consecutive series with the examiner: 1
Patient cannot perform three correct consecutive series even with the examiner: 0

#### 4. Conflicting instructions (sensitivity to interference)

"Tap twice when I tap once."

To ensure that the patient has understood the instruction, a series of 3 trials is run: 1-1-1.

Frontal assessment battery SVUH MedEl tool

1/2

"Tap once when I tap twice."

To ensure that the patient has understood the instruction, a series of 3 trials is run: 2-2-2.

The examiner then performs the following series: 1-1-2-1-2-2-1-1-2.

Score No errors: 3 1 -2 errors: 2 > 2 errors: 1

Patient taps like the examiner at least four consecutive times: 0

#### 5. Go-No Go (inhibitory control)

"Tap once when I tap once."

To ensure that the patient has understood the instruction, a series of 3 trials is run: 1-1-1.

"Do not tap when I tap twice."

To ensure that the patient has understood the instruction, a series of 3 trials is run: 2-2-2.

The examiner then performs the following series: 1-1-2-1-2-2-2-1-1-2.

Score No errors: 3 1 -2 errors: 2 > 2 errors: 1

Patient taps like the examiner at least four consecutive times: 0

#### 6. Prehension behaviour (environmental autonomy)

"Do not take my hands."

The examiner is seated in front of the patient. Place the patient's hands palm up on his knees. Without saying anything or looking at the patient, the examiner brings his own hands close to the patient's hands and touches the palms of both the patient's hands, to see if he will spontaneously take them. If the patient takes the examiner's hands, try again after asking the patient: "Now, do not take my hands."

#### Score

Patient does not take the examiner's hands: 3 Patient hesitates and asks what he/she has to do: 2

Patient takes the hands without hesitation: 1

Patient takes the examiner's hand even after he/she has been told not to do so: 0

#### Interpreting results

A cut off score of 12 on the FAB has a sensitivity of 77% and specificity of 87% in differentiating between frontal dysexecutive type dementias and DAT

#### ReferenceS

Dubois, B.; Litvan, I.; The FAB: A frontal assessment battery at bedside. Neurology. 55(11): 1621-1626, 2000.

Slachevsky, A; Dubois, B. Frontal Assessment Battery and Differential Diagnosis of Frontotemporal Dementia and Alzheimer Disease. Archives of Neurology. 61(7): 1104-1107, 2004.

#### **21.1.4** Tinetti

# TINETTI BALANCE ASSESSMENT TOOL

| Tinetti M | E, Williams | TF, Mayewski R, | Fall Risk | Index for | elderly pat | ients based | on number | of chronic dis- |
|---|---|---|---|---|---|---|---|---|
| abilities. | Am J Med | 1986:80:429-434 | | | | | | |

PATIENTS NAME \_\_\_\_\_ D.o.b. \_\_\_\_ Ward \_\_\_\_

#### BALANCE SECTION

Patient is seated in hard, armless chair;

| | | Date | | |
|---|---|---|---|---|
| Sitting Balance | Leans or slides in chair<br>Steady, safe | = 0<br>= 1 | | |
| Rises from chair | Unable to without help<br>Able, uses arms to help<br>Able without use of arms | = 0<br>= 1<br>= 2 | | |
| Attempts to rise | Unable to without help<br>Able, requires > 1 attempt<br>Able to rise, 1 attempt | = 0<br>= 1<br>= 2 | | |
| Immediate standing<br>Balance (first 5 seconds) | Unsteady (staggers, moves feet, trunk sway)<br>Steady but uses walker or other support<br>Steady without walker or other support | = 0<br>= 1<br>= 2 | | |
| Standing balance | Unsteady<br>Steady but wide stance and uses support<br>Narrow stance without support | = 0<br>= 1<br>= 2 | | |
| Nudged | Begins to fall<br>Staggers, grabs, catches self<br>Steady | = 0<br>= 1<br>= 2 | | |
| Eyes closed | Unsteady<br>Steady | = 0<br>= 1 | | |
| Turning 360 degrees | Discontinuous steps<br>Continuous | = 0<br>= 1 | | |
| Turining 500 degrees | Unsteady (grabs, staggers)<br>Steady | = 0<br>= 1 | | |
| Sitting down | Unsafe (misjudged distance, falls into chair)<br>Uses arms or not a smooth motion<br>Safe, smooth motion | = 0<br>= 1<br>= 2 | | |
| | Bala | nce score | /16 | /16 |

# TINETTI BALANCE ASSESSMENT TOOL

### GAIT SECTION

Patient stands with therapist, walks across room (+/- aids), first at usual pace, then at rapid pace.

| | | Date | | |
|---|---|---|---|---|
| Indication of gait<br>(Immediately after told to 'go'.) | Any hesitancy or multiple attempts<br>No hesitancy | = 0<br>= 1 | | |
| Step length and height | Step to<br>Step through R<br>Step through L | = 0<br>= 1<br>= 1 | | |
| Foot clearance | Foot drop<br>L foot clears floor<br>R foot clears floor | = 0<br>= 1<br>= 1 | | |
| Step symmetry | Right and left step length not equal<br>Right and left step length appear equal | = 0<br>= 1 | | |
| Step continuity | Stopping or discontinuity between steps<br>Steps appear continuous | = 0<br>= 1 | | |
| Path | Marked deviation<br>Mild/moderate deviation or uses w. aid<br>Straight without w. aid | = 0<br>= 1<br>= 2 | | |
| Trunk | Marked sway or uses w. aid<br>No sway but flex. knees or back or<br>uses arms for stability<br>No sway, flex., use of arms or w. aid | = 0<br>= 1<br>= 2 | | |
| Walking time | Heels apart<br>Heels almost touching while walking | = 0<br>= 1 | | |
| | | Gait score | /12 | /12 |
| | Balance score carried forward | | | |
| | Total Score = Balance + Gait score | | | |

#### Risk Indicators:

| Tinetti Tool Score | Risk of Falls |
|--------------------|---------------|
| ≤18 | High |
| 19-23 | Moderate |
| ≥24 | Low |

# 21.1.5 Addiction index in everyday activities (BADL)

| | Hygiene | Autonomous | 0 |
|---|------------|--------------------------------------------|---|
| | | Partial assistance for one part of | |
| | | the body | 1 |
| | | Assistance for several parts of the | |
| | | body or toileting impossible | 2 |
| | Dressing | Autonomous | 0 |
| | | Dresses but needs assistance with shoes | 1 |
| | | Needs assistance in choosing clothing, | |
| | | getting dressed, and remains partially | |
| | | or completely undressed | 2 |
| | Toileting | Autonomous | 0 |
| ľ | | Needs to be accompanied; needs | |
| | | assistance | 1 |
| | | Does not go to the toilet; does not use | |
| | | the toilet or urinal | 2 |
| | Locomotion | Autonomous | 0 |
| | | Needs assistance | 1 |
| | | Bedridden | 2 |
| | Continence | Continent | 0 |
| | | Occasionalincontinence | 1 |
| | | Permanentincontinence | 2 |
| | Meals | Autonomous | 0 |
| | | Needs assistance to cut meat or peel fruit | 1 |
| | | Total assistance or artificial feeding | 2 |
| | Total | | |

Version No.3 of 23.04.2018

Scale of Basic Activities of Daily Living (ADL)

# 21.1.6 Addiction index in the instrumental activities of daily life (IADL)

| Patient Name: | _ | Date: | |
|---|---|---|---|
| Patient ID # | _ | | |
| LAWTON - BRODY INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE (I.A.D.L.) | | | |
| Scoring: For each category, circle the item description that most closely resembles the client's highest functional level (either 0 or 1). | | | |
| A. Ability to Use Telephone | | E. Laundry | |
| 1. Operates telephone on own initiative-looks | 1 | Does personal laundry completely | 1 |
| up and dials numbers, etc. | | <ol><li>Launders small items-rinses stockings, etc.</li></ol> | 1 |
| 2. Dials a few well-known numbers | 1 | 3. All laundry must be done by others | 0 |
| <ol><li>Answers telephone but does not dial</li></ol> | 1 | | |
| 4. Does not use telephone at all | 0 | | |
| B. Shopping | | F. Mode of Transportation | |
| Takes care of all shopping needs independently | 1 | Travels independently on public transportation or<br>drives own car | 1 |
| 2. Shops independently for small purchases | 0 | <ol><li>Arranges own travel via taxi, but does not</li></ol> | 1 |
| <ol><li>Needs to be accompanied on any shopping</li></ol> | 0 | otherwise use public transportation | |
| trip | | 3. Travels on public transportation when | 1 |
| 4. Completely unable to shop | 0 | accompanied by another | |
| | | 4. Travel limited to taxi or automobile with | 0 |
| | | assistance of another | _ |
| 0.5.15 | _ | 5. Does not travel at all | 0 |
| C. Food Preparation | 1 | G. Responsibility for Own Medications | 1 |
| Plans, prepares and serves adequate meals independently | 1 | <ol> <li>Is responsible for taking medication in correct<br/>dosages at correct time</li> </ol> | 1 |
| 2. Prepares adequate meals if supplied with | 0 | Takes responsibility if medication is prepared in | 0 |
| ingredients | | advance in separate dosage | |
| 3. Heats, serves and prepares meals, or | 0 | 3. Is not capable of dispensing own medication | 0 |
| prepares meals, or prepares meals but does | | | |
| not maintain adequate diet | | | |
| 4. Needs to have meals prepared and served | 0 | | |
| D. Housekeeping | | H. Ability to Handle Finances | |
| Maintains house alone or with occasional | 1 | Manages financial matters independently | 1 |
| assistance (e.g. "heavy work domestic help") | ١. | (budgets, writes checks, pays rent, bills, goes to | |
| Performs light daily tasks such as dish | 1 | bank), collects and keeps track of income | |
| washing, bed making | ١, | Manages day-to-day purchases, but needs help | 1 |
| 3. Performs light daily tasks but cannot | 1 | with banking, major purchases, etc. | ^ |
| maintain acceptable level of cleanliness 4. Needs help with all home maintenance | 1 | 3. Incapable of handling money | 0 |
| tasks | 1 | | |
| 5. Does not participate in any housekeeping | 0 | | |
| tasks | ľ | | |
| Score | | Score | |
| | | Total score | |
| | | dent) to 8 (high function, independent) for women | |
| and 0 through 5 for men to avoid potential gende | er bias | S. | 1 |

# 21.1.7 Neuropsychiatric Inventory NPI-NH

| NPI-NH | Neuropsychiatric Inventory –<br>Nursing Home Version |
|--------|------------------------------------------------------|
| | Scoring Summary |

| Scoring Summary | | | | | | |
|---|---|---|---|---|---|---|
| CENTER# SCREENING# PATIENT # PATIENT INITIALS VISIT DATE | | | | | | |
| Please transcribe appropriate categories from the NPI-NH Worksheet into the boxes provided. | | | | | | |
| For each domain: - If symptoms of a domain did not apply, check the "N/A" box. - If symptoms of a domain were absent, check the "0" box. - If symptoms of a domain were present, check one score each for Frequency and Severity. - Multiply Frequency score x Severity score and enter the product in the space provided. - Total all Frequency x Severity scores and record the Total Score below. - If symptoms of a domain were present, check one score for Occupational Disruptiveness; total all occupational disruptiveness scores for a summary score. | | | | | | |
| DOMAIN | N/A <sup>1</sup> | ABSENT | FREQUENCY | SEVERITY | FREQUENCY<br>X SEVERITY | OCUPATIONAL<br>DISRUPTIVENESS |
| | | 0 | 1 2 3 4 | 1 2 3 | | 0 1 2 3 4 5 |
| A. Delusions | | | | | | |
| B. Hallucinations | | | | | | |

| DOMAIN | N/A1 | ABSENT | FREQUENCY | SEVERITY | FREQUENCY<br>X SEVERITY | OCUPATIONAL<br>DISRUPTIVENESS |
|---|---|---|---|---|---|---|
| | | 0 | 1 2 3 4 | 1 2 3 | | 0 1 2 3 4 5 |
| A. Delusions | | | | | | |
| B. Hallucinations | | | | | | |
| C. Agitation/Aggression | | | | | | 000000 |
| D. Depression/Dysphoria | | | | | | 000000 |
| E. Anxiety | | | | | | 000000 |
| F. Elation/Euphoria | | | | | | 000000 |
| G. Apathy/Indifference | | | | | | 000000 |
| H. Disinhibition | | | | | | 000000 |
| I. Irritability/Lability | | | | | | 000000 |
| J. Aberrant Motor Behavior | | | | | | 000000 |
| TOTAL SCORE: | | | | | | |
| K. Sleep and Nighttime<br>Behavior Disorders | | | | | | 000000 |
| L. Appetite/Eating Changes | | | | | | 000000 |

Version No.3 of 23.04.2018

# Neuropsychiatric Inventory -NPI-NH Nursing Home Version

# Worksheet

Directions: Read all items from the NPI-NH "Instructions for Administration of the NPI-NH". Mark Caregiver's responses on this worksheet before scoring the Frequency, Severity, and Occupational Disruptiveness.

| A. DELUSIONS: Yes No N/A Frequency Severity Occupational Disruptiveness 1. Fear of harm 2. Fear of theft 3. Spousal affair 4. Phantom boarder 5. Spouse imposter 6. House not home 7. Fear of abandonment 8. Talks to TV, etc. 9. Other | B. HALLUCINATIONS: Severity Occupational Disruptiveness 1. Hears voices 2. Talks to people not there 3. Sees things not there 4. Smells things not there 5. Feels things not there 6. Unusual taste sensations 7. Other |
|---|---|
| C. AGITATION/AGGRESSION: Frequency Severity Occupational Disruptiveness 1. Upset with caregiver; resists ADL's 2. Stubbornness 3. Uncooperative; resists help 4. Hard to handle 5. Cursing or shouting angrily 6. Slams doors; kicks, throws things 7. Hits, harms others 8. Other | D. DEPRESSION/DYSPHORIA: □Yes □No □N/A Frequency Severity Occupational Disruptiveness □ 1. Tearful and sobbing □ 2. States, acts as if sad □ 3. Puts self down, feels like failure □ 4. "Bad person", deserves punishment □ 5. Discouraged, no future □ 6. Burden to family □ 7. Talks about dying, killing self □ 8. Other |
| E. ANXIETY: Yes No N/A Frequency | F. ELATION/EUPHORIA: \( \text{ Yes } \) No \( \text{ N/A} \) Frequency Severity Occupational Disruptiveness \( \text{ 1. Feels too good, too happy} \) \( \text{ 2. Abnormal humor} \) \( \text{ 3. Childish, laughs inappropriately} \) \( \text{ 4. Jokes or remarks not funny to others} \) \( \text{ 5. Childish pranks} \) \( \text{ 6. Talks "big", grandiose} \) \( \text{ 7. Other} \) |

# Neuropsychiatric Inventory – NPI-NH Nursing Home Version

# Worksheet

| G. APATHY/INDIFFERENCE: Severity Occupational Disruptiveness 1. Less spontaneous or active 2. Less likely to initiate conversation 3. Less affectionate, lacking emotions 4. Contributes less to household chores 5. Less interested in others 6. Lost interest in friends or family 7. Less enthusiastic about interests 8. Other | H. DISINHIBITION: Yes No N/A FrequencySeverity Occupational Disruptiveness 1. Acts impulsively 2. Excessively familiar with strangers 3. Insensitive or hurtful remarks 4. Crude or sexual remarks 5. Talks openly of private matters 6. Inappropriate touching of others 7. Other |
|---|---|
| I. IRRITABILITY/LABILITY: Yes No N/A Frequency Severity Occupational Disruptiveness 1. Bad temper, "flies off handle" easily 2. Rapid changes in mood 3. Sudden flashes of anger 4. Impatient, trouble coping with delays 5. Cranky, irritable 6. Argues, difficult to get along with 7. Other | J. ABERRANT MOTOR BEHAVIOR: Frequency Severity Occupational Disruptiveness 1. Paces without purpose 2. Opens or unpacks closets or drawers 3. Repeatedly dresses and undresses 4. Repetitive activities or "habits" 5. Handling, picking, wrapping behavior 6. Excessively fidgety 7. Other |
| K. SLEEP AND NIGHTTIME BEHAVIOR DISORDERS: Yes No N/A Frequency Severity Occupational Disruptiveness 1. Difficulty falling asleep 2. Up during the night 3. Wanders, paces, inappropriate activity 4. Awakens others at night 5. Wakes and dresses to go out at night 6. Early morning awakening 7. Sleeps excessively during the day 8. Other | L. APPETITE/EATING CHANGES: Yes |

# 21.1.8 Clinical Dementia Rating (CDR)

| | Impairment | | | | |
|---|---|---|---|---|---|
| | None<br>0 | Questionable<br>0.5 | Mild<br>1 | Moderate<br>2 | Severe<br>3 |
| Memory | No memory loss or slight inconsistent forgetfulness | Consistent slight<br>forgetfulness; partial<br>recollection of events;<br>"benign" forgetfulness | Moderate memory loss;<br>more marked for recent<br>events; defect interferes<br>with everyday activities | Severe memory loss; only<br>highly learned material<br>retained; new material<br>rapidly lost | Severe memory loss;<br>only fragments remain |
| Orientation | Fully oriented | Fully oriented except for slight difficulty with time relationships | Moderate difficulty with<br>time relationships;<br>oriented for place at<br>examination; may have<br>geographic disorientation<br>elsewhere | Severe difficulty with time relationships; usually disoriented to time, often to place | Oriented to person only |
| Judgment & Problem<br>Solving | Solves everyday problems<br>& handles business &<br>financial affairs well;<br>judgment good in relation<br>to past performance | Slight impairment in<br>solving problems,<br>similarities, and<br>differences | Moderate difficulty in<br>handling problems,<br>similarities, and<br>differences; social<br>judgment usually<br>maintained | Severely impaired in<br>handling problems,<br>similarities, and<br>differences; social<br>judgment usually impaired | Unable to make judgments or solve problems |
| Community Affairs | Independent function at<br>usual level in job,<br>shopping, volunteer and<br>social groups | Slight impairment in these activities | Unable to function independently at these activities although may still be engaged in some; appears normal to casual inspection | No pretense of independent function outside home Appears well enough to be taken to functions outside a family home Appears too ill to be taken to functions outside a family home | |
| Home and Hobbies | Life at home, hobbies, and intellectual interests well maintained | Life at home, hobbies,<br>and intellectual interests<br>slightly impaired | Mild but definite<br>impairment of function at<br>home; more difficult<br>chores abandoned; more<br>complicated hobbies and<br>interests abandoned | Only simple chores<br>preserved; very restricted<br>interests, poorly<br>maintained | No significant function in home |
| Personal Care | Fully capable of self-care | | Needs prompting | Requires assistance in<br>dressing, hygiene,<br>keeping of personal<br>effects | Requires much help with<br>personal care; frequent<br>incontinence |

Score only as decline from previous usual level due to cognitive loss, not impairment due to other factors.